CLINICAL TRIAL: NCT03673904
Title: High Sensitive CRP Level in Prediabetics and Newly Diagnosed Type 2 Diabetic Patients
Brief Title: High Sensitive CRP in Prediabetics and Diabetes
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine, Fayoum University
Other Study IDs: D84
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Assess Level of High Sensitive CRP in Diabetics and Prediabetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prediabetics: Ages ranging from 18 to 60 years old,males and females were included . A fasting blood glucose level (100 to 125 mg/dL). or A 2-hour blood glucose level (140 to 199 mg/dL) .or Hb A1C 5.7% to 6.4%.
- Newly diagnosed type 2 diabetes: Ages ranging from 18 to 60 years old,males and females were included Newly diagnosed type 2 diabetes: (maximum within one month from diagnosis) A fasting blood glucose level >126 mg/dl A 2-hour blood glucose level > 200 mg/d Hb A1C > 6.5%

SUMMARY:
The aim of this study was to study the level of high-sensitivity CRP in sera of pre-diabetic and newly diagnosed patients with type 2 diabetes mellitus and its correlation with HOMA IR and HbA1c

DETAILED DESCRIPTION:
This study will include (180) subjects, 60 pre-diabetic patients, 60 patients with newly diagnosed type 2 diabetes ( within one month of diagnosis) and 60 normal healthy non diabetic individuals as a control group. The study individuals will be recruited from the Diabetes and Internal Medicine Clinics of Fayoum University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetic patients:

  * A fasting blood glucose level (100 to 125 mg/dL). or
  * A 2-hour blood glucose level (140 to 199 mg/dL) .or
  * Hb A1C 5.7% to 6.4%.
* Newly diagnosed type 2 diabetes: (maximum within one month from diagnosis)

  * A fasting blood glucose level >126 mg/dl
  * A 2-hour blood glucose level > 200 mg/dl
  * Hb A1C > 6.5%

Exclusion Criteria:

* Pregnant or lactating females.
* Patients who have recent infection.
* Patients with acute inflammatory diseases as autoimmune diseases.
* Patients with malignancy or on chemotherapy.
* Patients with acute or chronic liver or renal diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study individuals were recruited from the Diabetes and Internal Medicine Clinics of Fayoum University Hospital
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
statistical significant elevation of high sensitive CRP in diabetics and prediabetes | 2 years

IPD SHARING:
Plan to Share IPD: Undecided
still to be decided later